CLINICAL TRIAL: NCT02207231
Title: Phase 3, Multicenter, Randomized, Double-blind, Placebo and Active Comparator-controlled Study Evaluating the Efficacy and Safety of Guselkumab in the Treatment of Subjects With Moderate to Severe Plaque-type Psoriasis
Brief Title: A Study of Guselkumab in the Treatment of Participants With Moderate to Severe Plaque-Type Psoriasis
Acronym: VOYAGE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR105047; CNTO1959PSO3001 (Other: Janssen Research & Development, LLC); 2014-000719-15 (EudraCT Number)
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Psoriasis
Keywords: Psoriasis; Plaque-type psoriasis; Guselkumab; Adalimumab; CNTO 1959; Monoclonal antibody
MeSH Terms: conditions — Psoriasis | interventions — guselkumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental): Participants received Guselkumab 100 milligram (mg) at Weeks 0, 4, and 12 and every 8 weeks (q8w) thereafter through Week 252, placebo for guselkumab at Week 16, and placebo for adalimumab (two 0.8 milliliter [mL] injections) at Week 0 followed by one 0.8 mL injection at Weeks 1, 3, and 5, and every 2 weeks (q2w) thereafter through Week 47.
  Interventions: Drug: Guselkumab 100 mg; Drug: Placebo for guselkumab; Drug: Placebo for adalimumab
- Group II (Placebo Comparator): Participants received Placebo for guselkumab at Weeks 0, 4, and 12, and placebo for adalimumab (two 0.8 mL injections) at Week 0, followed by one 0.8 mL injection at Weeks 1, 3, and 5, and q2w through Week 15. At Week 16, placebo participants will cross over to receive guselkumab 100 mg at Weeks 16 and 20 and q8w thereafter through Week 252, as well as placebo for adalimumab at Weeks 17, 19, 21, and 23, and q2w thereafter through Week 47.
  Interventions: Drug: Guselkumab 100 mg; Drug: Placebo for guselkumab; Drug: Placebo for adalimumab
- Group III (Active Comparator): Participants received Adalimumab 80 mg at Week 0 (two 40 mg [0.8 mL] injections) and 40 mg at Weeks 1, 3, 5, and q2w thereafter through Week 47, placebo for guselkumab at Weeks 0, 4, 12, 16, and 20, and q8w thereafter through Week 44 and guselkumab 100 mg at Weeks 52, 60, and q8w thereafter through Week 252.
  Interventions: Drug: Guselkumab 100 mg; Drug: Placebo for guselkumab; Drug: Adalimumab

INTERVENTIONS:
Drug: Guselkumab 100 mg — 100 mg by subcutaneous injection at Weeks 0, 4 and q8w thereafter through Week 252 (Group 1). 100 mg by subcutaneous injection at Weeks 16, 20 and q8w thereafter through Week 252 (Group II). 100 mg by subcutaneous injection at Week 52 and q8w thereafter through Week 252 (Group III).
  Other Names: CNTO 1959
Drug: Placebo for guselkumab — Subcutaneous injections to maintain the blind.
Drug: Adalimumab — 80 mg by subcutaneous injection at Week 0, then 40 mg at Week 1 and every 2 weeks (q2w) thereafter through Week 47.
  Other Names: HUMIRA®
  Arms: Group III
Drug: Placebo for adalimumab — Subcutaneous injections to maintain the blind.
  Arms: Group I; Group II

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of guselkumab (CNTO 1959) in the treatment of participants with moderate to severe plaque-type psoriasis.

DETAILED DESCRIPTION:
This is a randomized (assignment of study drug by chance), double-blind (neither the participant or study staff will know the identity of study drugs), placebo- (inactive substance identical in appearance to study drug) and active-comparator-controlled (use of an approved drug to compare with study drug) study of guselkumab in participants with moderate to severe plaque-type psoriasis (scaly skin rash). The active comparator study drug is adalimumab, an approved drug for the treatment of moderate to severe plaque psoriasis. Participants who satisfy all inclusion and exclusion criteria will be randomly assigned in a 2:1:2 ratio to one of three treatment groups (arms): Group I (guselkumab 100 mg dose regimen), Group II (placebo then crossover to guselkumab at Week 16), or Group III (adalimumab at standard psoriasis dosing). All participants will receive guselkumab every 8 weeks (q8w) from Week 52 through Week 252 (open label treatment period).The end of the study is defined as the time the last participant completes the Week 264 visit. Participants will primarily be assessed for Investigator's Global Assessment (IGA) Score of 0 or 1 and Psoriasis Area and Severity Index (PASI) 90 Response at Week 16. The total duration of the study will be approximately 268 weeks (includes a 4-week screening period). Participants will be monitored for safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of plaque-type psoriasis (with or without psoriatic arthritis) at least 6 months before the first administration of study agent
* Have a Psoriasis Area and Severity Index (PASI) greater than or equal to (>=) 12 at Screening and at Baseline
* Have an Investigator's Global Assessment (IGA) score >=3 at Screening and at Baseline
* Have an involved body surface area (BSA) >=10 percent (%) at Screening and at Baseline
* Must be a candidate for either systemic therapy or phototherapy for psoriasis

Exclusion Criteria:

* Participants with nonplaque forms of psoriasis (for example, erythrodermic, guttate, or pustular) or with current drug-induced psoriasis (for example, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* Participants who have ever received guselkumab or adalimumab
* History or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Has any condition that, in the opinion of the investigator, would make participation not be in the best interest (for example, compromise the well-being) of the participant or that could prevent, limit, or confound the protocol-specified assessments
* Is pregnant, nursing, or planning a pregnancy (both men and women) within 5 months following the last administration of study drug

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 837 (Actual)
Dates: Start 2014-11-26 (Actual); Primary Completion 2015-09-29 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (97):
- United States (26):
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Farmington, Connecticut
  - Clearwater, Florida
  - Coral Gables, Florida
  - Ocala, Florida
  - Alpharetta, Georgia
  - Rolling Meadows, Illinois
  - Plainfield, Indiana
  - Boston, Massachusetts
  - Troy, Michigan
  - New Brighton, Minnesota
  - St Louis, Missouri
  - East Windsor, New Jersey
  - Albuquerque, New Mexico
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Johnston, Rhode Island
  - Arlington, Texas
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Webster, Texas
  - Norfolk, Virginia
- Australia (8):
  - Darlinghurst
  - East Melbourne
  - Hectorville
  - Liverpool
  - Melbourne
  - Westmead
  - Woden
  - Woolloongabba
- Canada (10):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Ajax, Ontario
  - London, Ontario
  - North Bay, Ontario
  - Peterborough, Ontario
  - Montreal, Quebec
- Germany (12):
  - Berlin
  - Bonn
  - Dresden
  - Essen
  - Frankfurt am Main
  - Gera
  - Hamburg
  - Kiel
  - Lübeck
  - Mahlow
  - Münster
  - Tübingen
- Hungary (6):
  - Budapest
  - Debrecen
  - Kaposvár
  - Kecskemét
  - Pécs
  - Szeged
- Poland (6):
  - Bialystok
  - Bydgoszcz
  - Lodz
  - Olsztyn
  - Warsaw
  - Wroclaw
- Russia (10):
  - Kirov
  - Krasnodar
  - Lipetsk
  - Moscow
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Stavropol
  - Ulyanovsk
  - Yekaterinburg
- South Korea (5):
  - Bundang
  - Busan
  - Daejeon
  - Seoul
  - Suwon
- Spain (9):
  - Barakaldo
  - Barcelona
  - Córdoba
  - Madrid
  - Manises
  - Palma de Mallorca
  - Salamanca
  - San Sebastián de los Reyes
  - Valencia
- Taiwan (5):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District

REFERENCES:
- [Derived] Puig L, Costanzo A, de Jong EMGJ, Torres T, Warren RB, Wapenaar R, Wegner S, Gorecki P, Gramiccia T, Jazra M, Buyze J, Conrad C. Progression of Quality of Life in Patients with Plaque Psoriasis Who Achieved Three or More Years of Complete Skin Clearance with Guselkumab Treatment: a Post hoc Analysis of the VOYAGE 1 Clinical Trial. Dermatol Ther (Heidelb). 2024 Sep;14(9):2539-2558. doi: 10.1007/s13555-024-01245-6. Epub 2024 Aug 17. PMID 39153060
- [Derived] Blauvelt A, Langley RG, Branigan PJ, Liu X, Chen Y, DePrimo S, Ma K, Scott B, Campbell K, Munoz-Elias EJ, Papp KA. Guselkumab Reduces Disease- and Mechanism-Related Biomarkers More Than Adalimumab in Patients with Psoriasis: A VOYAGE 1 Substudy. JID Innov. 2024 Jun 5;4(5):100287. doi: 10.1016/j.xjidi.2024.100287. eCollection 2024 Sep. PMID 39114670
- [Derived] Egeberg A, Conrad C, Gorecki P, Wegner S, Buyze J, Acciarri L, Thaci D. Response Types and Factors Associated with Response Types to Biologic Therapies in Patients with Moderate-to-Severe Plaque Psoriasis from Two Randomized Clinical Trials. Dermatol Ther (Heidelb). 2024 Mar;14(3):745-758. doi: 10.1007/s13555-024-01123-1. Epub 2024 Mar 15. PMID 38485863
- [Derived] Strober B, Coates LC, Lebwohl MG, Deodhar A, Leibowitz E, Rowland K, Kollmeier AP, Miller M, Wang Y, Li S, Chakravarty SD, Chan D, Shawi M, Yang YW, Thaҫi D, Rahman P. Long-Term Safety of Guselkumab in Patients with Psoriatic Disease: An Integrated Analysis of Eleven Phase II/III Clinical Studies in Psoriasis and Psoriatic Arthritis. Drug Saf. 2024 Jan;47(1):39-57. doi: 10.1007/s40264-023-01361-w. Epub 2023 Oct 31. PMID 37906417
- [Derived] Puig L, Costanzo A, de Jong EMGJ, Torres T, Warren RB, Wapenaar R, Wegner S, Gorecki P, Gramiccia T, Jazra M, Buyze J, Conrad C. Guselkumab-Treated Patients with Plaque Psoriasis Who Achieved Complete Skin Clearance for >/= 156 Consecutive Weeks: A Post-Hoc Analysis From the VOYAGE 1 Clinical Trial. Am J Clin Dermatol. 2024 Mar;25(2):315-325. doi: 10.1007/s40257-023-00816-1. Epub 2023 Oct 7. PMID 37804472
- [Derived] Kim BS, Jo SJ, Youn S, Reich K, Saadoun C, Chang CL, Yang YW, Huang YH, Tsai TF. Five-year Maintenance of Clinical Response and Consistent Safety Profile for Guselkumab in Asian patients with Psoriasis from VOYAGE 1 and VOYAGE 2. Dermatol Ther (Heidelb). 2023 Nov;13(11):2721-2737. doi: 10.1007/s13555-023-01026-7. Epub 2023 Sep 26. PMID 37750995
- [Derived] Orbai AM, Chakravarty SD, You Y, Shawi M, Yang YW, Merola JF. Efficacy of Guselkumab in Treating Nails, Scalp, Hands, and Feet in Patients with Psoriasis and Self-reported Psoriatic Arthritis. Dermatol Ther (Heidelb). 2023 Nov;13(11):2859-2868. doi: 10.1007/s13555-023-01012-z. Epub 2023 Sep 15. PMID 37713133
- [Derived] Reich K, Gordon KB, Strober BE, Armstrong AW, Miller M, Shen YK, You Y, Han C, Yang YW, Foley P, Griffiths CEM. Five-year maintenance of clinical response and health-related quality of life improvements in patients with moderate-to-severe psoriasis treated with guselkumab: results from VOYAGE 1 and VOYAGE 2. Br J Dermatol. 2021 Dec;185(6):1146-1159. doi: 10.1111/bjd.20568. Epub 2021 Sep 8. PMID 34105767
- [Derived] Armstrong AW, Reich K, Foley P, Han C, Song M, Shen YK, You Y, Papp KA. Improvement in Patient-Reported Outcomes (Dermatology Life Quality Index and the Psoriasis Symptoms and Signs Diary) with Guselkumab in Moderate-to-Severe Plaque Psoriasis: Results from the Phase III VOYAGE 1 and VOYAGE 2 Studies. Am J Clin Dermatol. 2019 Feb;20(1):155-164. doi: 10.1007/s40257-018-0396-z. PMID 30417277
- [Derived] Foley P, Gordon K, Griffiths CEM, Wasfi Y, Randazzo B, Song M, Li S, Shen YK, Blauvelt A. Efficacy of Guselkumab Compared With Adalimumab and Placebo for Psoriasis in Specific Body Regions: A Secondary Analysis of 2 Randomized Clinical Trials. JAMA Dermatol. 2018 Jun 1;154(6):676-683. doi: 10.1001/jamadermatol.2018.0793. PMID 29799960

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Guselkumab 100 mg: Participants received placebo matched to guselkumab subcutaneous injection at Weeks 0, 4, and 12, and placebo matched to adalimumab (2 subcutaneous injections) at Week 0, followed by placebo matched to adalimumab (1 subcutaneous injection) at Weeks 1, 3, and 5 and once every 2 weeks thereafter through Week 15 in the placebo controlled period (PCP). Participants then crossed over to receive guselkumab 100 milligram (mg) subcutaneous injection at Weeks 16 and 20 and once every 8 weeks thereafter through Week 44 and placebo matched to adalimumab subcutaneous injection at Weeks 17, 19, 21, and 23 and every 2 weeks thereafter through Week 47 in the active controlled period (ACP). Participants continued to receive guselkumab 100 mg subcutaneously q8w at Week 52 and thereafter through Week 252 in the open-label treatment period.
- Guselkumab 100 mg: Participants received guselkumab 100 mg subcutaneous injection at Weeks 0, 4, and 12 and once every 8 weeks thereafter through Week 44, placebo matched to guselkumab subcutaneous injection at Week 16, and placebo matched to adalimumab (2 subcutaneous injections) at Week 0 followed by placebo matched to adalimumab (1 subcutaneous injection) at Weeks 1, 3, and 5 and every 2 weeks thereafter through Week 47. Participants receiving guselkumab continued to receive guselkumab 100mg subcutaneously q8w at Week 52 and thereafter through Week 252 in the open label period.
- Adalimumab Then Guselkumab 100 mg: Participants received adalimumab 80 mg (2 subcutaneous injections) at Week 0 and adalimumab 40 mg (1 subcutaneous injection) at Weeks 1, 3, 5 and once every 2 weeks thereafter through Week 47 and placebo matched to guselkumab subcutaneous injection at Weeks 0, 4, 12, 16, 20 and once every 8 weeks thereafter through Week 44. Participants entered a washout period after their final dose of adalimumab at Week 47 and received guselkumab 100 mg subcutaneously q8w at Week 52 and thereafter through Week 252.
- Guselkumab Combined: All participants who received guselkumab 100 mg subcutaneously q8w at Week 52 and thereafter through Week 252.
Period: Placebo Controlled Period: Week 0 - 16
Arm/Group | Placebo Then Guselkumab 100 mg | Guselkumab 100 mg | Adalimumab Then Guselkumab 100 mg | Guselkumab Combined
Started | 174 | 329 | 334 | 0
Treated | 174 | 329 | 333 | 0
Completed | 167 | 322 | 324 | 0
Not Completed | 7 | 7 | 10 | 0
Not completed — Adverse Event | 2 | 4 | 2 | 0
Not completed — Lack of Efficacy | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 4 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Noncompliance | 0 | 2 | 1 | 0
Period: Active Controlled Period: Week 16 - 48
Arm/Group | Placebo Then Guselkumab 100 mg | Guselkumab 100 mg | Adalimumab Then Guselkumab 100 mg | Guselkumab Combined
Started | 165 (2 participants did not cross-over.) | 322 | 324 | 0
Completed | 162 | 301 | 281 | 0
Not Completed | 3 | 21 | 43 | 0
Not completed — Adverse Event | 1 | 6 | 10 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 3 | 11 | 0
Not completed — Lost to Follow-up | 1 | 2 | 5 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 10 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Noncompliance | 0 | 3 | 3 | 0
Not completed — Other | 0 | 2 | 3 | 0
Period: Open-label Guselkumab: Week 48 - 264
Arm/Group | Placebo Then Guselkumab 100 mg | Guselkumab 100 mg | Adalimumab Then Guselkumab 100 mg | Guselkumab Combined
Started | 0 | 0 | 280 (One participant did not crossover at Week 52 due to adverse event.) | 463 (162 + 301= 463)
Completed | 0 | 0 | 242 | 380
Not Completed | 0 | 0 | 38 | 83
Not completed — Adverse Event | 0 | 0 | 12 | 19
Not completed — Death | 0 | 0 | 1 | 3
Not completed — Pregnancy | 0 | 0 | 3 | 7
Not completed — Lack of Efficacy | 0 | 0 | 2 | 4
Not completed — Lost to Follow-up | 0 | 0 | 6 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 10 | 28
Not completed — Other | 0 | 0 | 4 | 11

BASELINE CHARACTERISTICS:
Population: Randomized analysis set included all participants who were randomized at Week 0.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Guselkumab 100 mg | Guselkumab 100 mg | Adalimumab Then Guselkumab 100 mg | Total
Number analyzed (Participants) | 174 | 329 | 334 | 837
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 3 | 3
  Between 18 and 65 years | 164 | 311 | 315 | 790
  >=65 years | 10 | 18 | 16 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (12.9) | 43.9 (12.74) | 42.9 (12.58) | 43.7 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 89 | 85 | 229
  Male | 119 | 240 | 249 | 608
Region of Enrollment [Number; unit: participants]
  Australia | 13 | 23 | 21 | 57
  Taiwan, Province Of China | 15 | 31 | 27 | 73
  Hungary | 7 | 9 | 14 | 30
  Poland | 22 | 42 | 43 | 107
  Russia | 21 | 48 | 49 | 118
  Canada | 24 | 50 | 48 | 122
  United States | 38 | 65 | 67 | 170
  Germany | 23 | 41 | 43 | 107
  Spain | 4 | 8 | 13 | 25
  Korea, Democratic People'S Republic Of | 7 | 12 | 9 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) in the Guselkumab Group Compared to the Placebo Group at Week 16
Description: The IGA documents the investigator's assessment of the participants' psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participants' psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Time Frame: Week 16
Population: Randomized analysis set include all participants randomized at Week 0. Nonresponder imputation (participants who met treatment-failure criteria before Week 16 or who did not come for evaluation at week 16 were considered nonresponders) was used to impute missing values.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received placebo matched to guselkumab subcutaneous injection at Weeks 0, 4, and 12, and placebo matched to adalimumab (2 subcutaneous injections) at Week 0, followed by placebo matched to adalimumab (1 subcutaneous injection) at Weeks 1, 3, and 5 and once every 2 weeks thereafter through Week 15 in the placebo controlled period (PCP).
- Guselkumab: Participants received guselkumab 100 mg subcutaneous injection at Weeks 0, 4, and 12 and placebo matched to adalimumab (2 subcutaneous injections) at Week 0 followed by placebo matched to adalimumab (1 subcutaneous injection) at Weeks 1, 3, and 5 and every 2 weeks thereafter through Week 15.
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 174 | 329
percentage of participants | 6.9 | 85.1
Statistical Analysis 1: Comparison: Placebo vs Guselkumab; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

2. Primary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index (PASI) 90 Response in the Guselkumab Group Compared to the Placebo Group at Week 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 percent improvement from baseline in the PASI score.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 174 | 329
percentage of participants | 2.9 | 73.3
Statistical Analysis 1: Comparison: Placebo vs Guselkumab; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

3. Secondary Outcome: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score of Cleared (0) in the Guselkumab Group Compared to the Adalimumab Group at Week 24 and 48
Description: as for outcome 1
Time Frame: Week 24 and 48
Population: Randomized analysis set included all participants randomized at Week 0. Nonresponder imputation (participants who met treatment-failure criteria before Week 24 or Week 48 or who did not come for evaluation at Week 24 or Week 48 were considered nonresponders, respectively, for Week 24 or Week 48 outcome measures) was used to impute missing values.
Measure: Number; unit: percentage of participants
Groups:
- Guselkumab: Participants received guselkumab 100 mg subcutaneous injection at Weeks 0, 4, and 12 and once every 8 weeks thereafter through Week 44, placebo matched to guselkumab subcutaneous injection at Week 16, and placebo matched to adalimumab (2 subcutaneous injections) at Week 0 followed by placebo matched to adalimumab (1 subcutaneous injection) at Weeks 1, 3, and 5 and every 2 weeks thereafter through Week 47.
- Adalimumab: Participants received adalimumab 80 mg (2 subcutaneous injections) at Week 0 and adalimumab 40 mg (1 subcutaneous injection) at Weeks 1, 3, 5 and once every 2 weeks thereafter through Week 47 and placebo matched to guselkumab subcutaneous injection at Weeks 0, 4, 12, 16, 20 and once every 8 weeks thereafter through Week 44.
Arm/Group | Guselkumab | Adalimumab
Number analyzed (Participants) | 329 | 334
percentage of participants
  Week 24 | 52.6 | 29.3
  Week 48 | 50.5 | 25.7
Statistical Analysis 1: Comparison: Guselkumab vs Adalimumab; Week 24; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test
Statistical Analysis 2: Comparison: Guselkumab vs Adalimumab; Week 48; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

4. Secondary Outcome: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) in the Guselkumab Group Compared to the Adalimumab Group at Week 24 and 48
Description: as for outcome 1
Time Frame: Week 24 and 48
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab | Adalimumab
Number analyzed (Participants) | 329 | 334
percentage of participants
  Week 24 | 84.2 | 61.7
  Week 48 | 80.5 | 55.4
Statistical Analysis 1: Comparison: Guselkumab vs Adalimumab; Week 24; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test
Statistical Analysis 2: Comparison: Guselkumab vs Adalimumab; Week 48; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

5. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index (PASI) 90 Response in the Guselkumab Group Compared to the Adalimumab Group at Week 24 and 48
Description: as for outcome 2
Time Frame: Week 24 and 48
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab | Adalimumab
Number analyzed (Participants) | 329 | 334
percentage of participants
  Week 24 | 80.2 | 53.0
  Week 48 | 76.3 | 47.9
Statistical Analysis 1: Comparison: Guselkumab vs Adalimumab; Week 24; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test
Statistical Analysis 2: Comparison: Guselkumab vs Adalimumab; Week 48; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

6. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Week 16 in the Guselkumab Group Compared to the Placebo Group
Description: The DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The DLQI total score ranges from 0 (not at all) to 30 (very much): 0-1 = no effect at all on the participant's life; 2-6 = small effect on the participant's life; 7-12 = moderate effect on the participant's life; 13-18 = very large effect on the participant's life; 19-30 = extremely large effect on the participant's life. Higher scores indicate more impact on quality of life of participants. This secondary outcome measure was planned to include only the placebo and guselkumab arms.
Time Frame: Baseline, Week 16
Population: Randomized analysis set included all participants who were randomized at Week 0 and have a baseline DLQI score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 174 | 329
units on a scale | -0.6 (6.36) | -11.2 (7.24)
Statistical Analysis 1: Comparison: Placebo vs Guselkumab; p value is based on analysis of variance (ANOVA) model stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, ANOVA

7. Secondary Outcome: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) in the Guselkumab Group Compared to the Adalimumab Group at Week 16
Description: as for outcome 1
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Adalimumab: Participants received adalimumab 80 mg (2 subcutaneous injections) at Week 0 and adalimumab 40 mg (1 subcutaneous injection) at Weeks 1, 3, 5 and once every 2 weeks thereafter through Week 15 and placebo matched to guselkumab subcutaneous injection at Weeks 0, 4, and 12.
Arm/Group | Guselkumab | Adalimumab
Number analyzed (Participants) | 329 | 334
percentage of participants | 85.1 | 65.9
Statistical Analysis 1: Comparison: Guselkumab vs Adalimumab; p value is based on 1-sided Mantel Haenszel (MH) Z-test adjusted for investigator site (pooled); Test type: Non-Inferiority or Equivalence — non-inferiority margin= 10.0%; p < 0.001, MH Z-test; Difference in Percentage = 19.3, 95% CI 2-sided [12.9 to 25.7]
Statistical Analysis 2: Comparison: Guselkumab vs Adalimumab; p value is based on the Cochran-Mantel-Haenszel chi-square test stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

8. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index (PASI) 90 Response in the Guselkumab Group Compared to the Adalimumab Group at Week 16
Description: as for outcome 2
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab | Adalimumab
Number analyzed (Participants) | 329 | 334
percentage of participants | 73.3 | 49.7
Statistical Analysis 1: Comparison: Guselkumab vs Adalimumab; p value is based on 1-sided MH Z-test adjusted for investigator site (pooled); Test type: Non-Inferiority or Equivalence — non-inferiority margin= 10.0%; p < 0.001, MH Z-test; Difference in Percentage = 24.1, 95% CI 2-sided [17.0 to 31.0]
Statistical Analysis 2: Comparison: Guselkumab vs Adalimumab; p value is based on the Cochran-Mantel-Haenszel chi-square test stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

9. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index (PASI) 75 Response in the Guselkumab Group Compared to the Adalimumab Group at Week 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 75 response represents participants who achieved at least a 75 percent improvement from baseline in the PASI score.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab | Adalimumab
Number analyzed (Participants) | 329 | 334
percentage of participants | 91.2 | 73.1
Statistical Analysis 1: Comparison: Guselkumab vs Adalimumab; p value is based on 1-sided MH Z-test adjusted for investigator site (pooled); Test type: Non-Inferiority or Equivalence — non-inferiority margin= 10%; p < 0.001, MH Z-test; Difference in percentage = 18.0, 95% CI 2-sided [12.4 to 23.8]
Statistical Analysis 2: Comparison: Guselkumab vs Adalimumab; p value is based on the Cochran-Mantel-Haenszel chi-square test stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

10. Secondary Outcome: Percentage of Participants Who Achieved a Scalp-specific Investigator's Global Assessment (Ss-IGA) Score of 0 or 1 and at Least a 2-Grade Improvement From Baseline at Week 16 in the Guselkumab Group Compared to the Placebo Group
Description: The ss-IGA instrument is used to evaluate the disease severity of scalp psoriasis. The lesions were assessed in terms of the clinical signs of redness, thickness, and scaliness, which are scored on a 5-point scale ranging from 0 = absence of disease, 1 = very mild disease, 2 = mild disease, 3 = moderate disease, and 4 = severe disease. This secondary outcome measure was planned to include only the placebo and guselkumab arms.
Time Frame: Week 16
Population: Population analyzed included only randomized participants at Week 0 who had an ss-IGA score greater than or equal to (>=) 2 at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 145 | 277
percentage of participants | 14.5 | 83.4
Statistical Analysis 1: Comparison: Placebo vs Guselkumab; p value is based on the Cochran-Mantel-Haenszel chi-square test stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

11. Secondary Outcome: Change From Baseline in Psoriasis Symptom and Sign Diary (PSSD) Symptom Score at Week 16 in the Guselkumab Group Compared to the Placebo Group
Description: The PSSD (24-hour version) is a patient-reported outcome (PRO) questionnaire designed and validated to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. It consisted of 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 (absent) to 10 (worst imaginable) numerical rating scales for severity. Items were averaged on the daily symptom score and sign score when at least 3 items (>=50 percentage of 5 items) on these scales are answered. The average value is converted into 0-100 scoring, such that Symptom [or Sign] score = average value*10, where, 0= least severe and 100= most severe and higher score indicates more severe disease. This secondary outcome measure was planned to include only the placebo and guselkumab arms.
Time Frame: Baseline and Week 16
Population: PSSD analysis set included all those participants who had baseline PSSD scores as the average score of at least 4 days out of the 7 days prior to the Week 0 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 129 | 249
units on a scale | -3.0 (19.56) | -41.9 (24.61)
Statistical Analysis 1: Comparison: Placebo vs Guselkumab; p value is based on ANOVA model stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, ANOVA

12. Secondary Outcome: Percentage of Participants Who Achieved a Psoriasis Symptom and Sign Diary (PSSD) Symptom Score of 0 in the Guselkumab Group Compared to the Adalimumab Group at Week 24
Description: The PSSD (24-hour version) is a patient-reported outcome (PRO) questionnaire designed and validated to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. It consisted of 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 (absent) to 10 (worst imaginable) numerical rating scales for severity. Items were averaged on the daily symptom score and sign score when at least 3 items (>=50 percentage of 5 items) on these scales are answered. The average value is converted into 0-100 scoring, such that Symptom [or Sign] score = average value*10, where, 0= least severe and 100= most severe and higher score indicates more severe disease.
Time Frame: Week 24
Population: PSSD analysis set included all those participants who were randomized at Week 0 and had baseline PSSD score greater than 0.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab | Adalimumab
Number analyzed (Participants) | 248 | 273
percentage of participants | 36.3 | 21.6
Statistical Analysis 1: Comparison: Guselkumab vs Adalimumab; p value is based on the Cochran-Mantel-Haenszel chi-square test stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

13. Secondary Outcome: Percentage of Participants Who Achieved PASI 90 Response at Week 252
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 percent improvement from baseline in the PASI score. As per planned analysis, participants from the baseline guselkumab group and the placebo crossover group were combined into a single guselkumab group for assessment of this outcome measure.
Time Frame: Week 252
Population: Population analyzed included participants who were randomized at Week 0 and treated with guselkumab. The analysis was performed using observed data after applying treatment failure rules. Here, N (Number of participants analyzed) signifies participants who were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- Guselkumab Combined: All participants who crossed over to receive guselkumab 100 mg subcutaneously at Week 16 from placebo group and participants who were randomized to guselkumab 100 mg group at Week 0. Placebo crossover participants were included in the guselkumab column after crossover to guselkumab.
Arm/Group | Guselkumab Combined | Adalimumab Then Guselkumab 100 mg
Number analyzed (Participants) | 391 | 246
percentage of participants | 84.1 | 82.5

14. Secondary Outcome: Percentage of Participants Who Achieved PASI 75 Response at Week 252
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 75 response represents participants who achieved at least a 75 percent improvement from baseline in the PASI score. As per planned analysis, participants from the baseline guselkumab group and the placebo crossover group were combined into a single guselkumab group for assessment of this outcome measure.
Time Frame: Week 252
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab Combined | Adalimumab Then Guselkumab 100 mg
Number analyzed (Participants) | 391 | 246
percentage of participants | 93.9 | 93.1

15. Secondary Outcome: Percentage of Participants Who Achieved an IGA Score of Cleared (0) or Minimal (1) at Week 252
Description: The IGA documents the investigator's assessment of the participants' psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participants' psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4). As per planned analysis, participants from the baseline guselkumab group and the placebo crossover group were combined into a single guselkumab group for assessment of this outcome measure.
Time Frame: Week 252
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab Combined | Adalimumab Then Guselkumab 100 mg
Number analyzed (Participants) | 391 | 246
percentage of participants | 82.4 | 82.9

16. Secondary Outcome: Percentage of Participants With a DLQI Score of 0 or 1 at Week 252
Description: The DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The DLQI total score ranges from 0 (not at all) to 30 (very much): 0-1 = no effect at all on the participant's life; 2-6 = small effect on the participant's life; 7-12 = moderate effect on the participant's life; 13-18 = very large effect on the participant's life; 19-30 = extremely large effect on the participant's life. Higher scores indicate more impact on quality of life of participants. As per planned analysis, participants from the baseline guselkumab group and the placebo crossover group were combined into a single guselkumab group for assessment of this outcome measure.
Time Frame: Week 252
Population: Population analyzed included participants who were randomized at Week 0 and treated with guselkumab with baseline DLQI score >1. The analysis was performed using observed data after applying treatment failure rules. Here, N (Number of participants analyzed) signifies participants who were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab Combined | Adalimumab Then Guselkumab 100 mg
Number analyzed (Participants) | 374 | 235
percentage of participants | 72.7 | 74.0

17. Secondary Outcome: Percentage of Participants Who Achieved a PSSD Symptom Score of 0 at Week 252
Description: The PSSD (24-hour version) is a PRO questionnaire designed and validated to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. It consisted of 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 (absent) to 10 (worst imaginable) numerical rating scales for severity. Items were averaged on the daily symptom score and sign score when at least 3 items (>=50 percentage of 5 items) on these scales are answered. The average value is converted into 0-100 scoring, such that Symptom score = average value*10, where, 0= least severe and 100= most severe and higher score indicates more severe disease. As per planned analysis, participants from the baseline guselkumab group and the placebo crossover group were combined into a single guselkumab group for assessment of this outcome measure.
Time Frame: Week 252
Population: Population analyzed included participants who were randomized at Week 0 and treated with guselkumab with baseline PSSD symptom score >0. The analysis was performed using observed data after applying treatment failure rules. Here, N (Number of participants analyzed) signifies participants who were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab Combined | Adalimumab Then Guselkumab 100 mg
Number analyzed (Participants) | 297 | 200
percentage of participants | 42.4 | 48.0

18. Secondary Outcome: Percentage of Participants Who Achieved a PSSD Sign Score of 0 at Week 252
Description: The PSSD (24-hour version) is a PRO questionnaire designed and validated to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. It consisted of 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 (absent) to 10 (worst imaginable) numerical rating scales for severity. Items were averaged on the daily symptom score and sign score when at least 3 items (>=50 percentage of 5 items) on these scales are answered. The average value is converted into 0-100 scoring, such that Sign score = average value*10, where, 0= least severe and 100= most severe and higher score indicates more severe disease. As per planned analysis, participants from the baseline guselkumab group and the placebo crossover group were combined into a single guselkumab group for assessment of this outcome measure.
Time Frame: Week 252
Population: Population analyzed included participants who were randomized at Week 0 and treated with guselkumab with baseline PSSD sign score >0. The analysis was performed using observed data after applying treatment failure rules. Here, N (Number of participants analyzed) signifies participants who were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab Combined | Adalimumab Then Guselkumab 100 mg
Number analyzed (Participants) | 297 | 201
percentage of participants | 33.0 | 37.8

ADVERSE EVENTS:
Time Frame: Baseline (Week 0) up to Week 264
Description: Safety analysis- participants who were randomized at Week 0, received at least 1 dose of study drug (partial/complete). Participants who discontinued treatment prematurely were followed for at least 12 weeks after last dose. Participants who discontinued in 1st period and had safety follow-up beyond Week 16, counted in both periods for safety. Discrepancy in number of participants in participant flow and numbers at risk in adverse events for GUS combined arm is justified in GUS arm description.
Groups:
- Placebo (PCP): Participants received placebo matched to guselkumab subcutaneous injection at Weeks 0, 4, and 12 during the placebo controlled period.
- Guselkumab 100 mg (PCP): Participants received guselkumab 100 mg subcutaneous injection at Weeks 0, 4, and 12 during the placebo controlled period.
- Adalimumab (PCP): Participants received adalimumab 80 mg (2 subcutaneous injections) at Week 0 and adalimumab 40 mg (1 subcutaneous injection) at Week 1 and once every other week thereafter through Week 15 during the placebo controlled period.
- Placebo Then Guselkumab 100 mg (ACP): Participants initially randomized to placebo crossed over to receive guselkumab 100 milligram (mg) subcutaneous injection at Weeks 16 and 20 and once every 8 weeks thereafter through Week 44 in the active controlled period (ACP).
- Guselkumab 100 mg (ACP): Participants received guselkumab 100 mg subcutaneous injection at Weeks 0, 4, and 12 and once every 8 weeks thereafter through Week 44, placebo matched to guselkumab subcutaneous injection at Week 16, and placebo matched to adalimumab (2 subcutaneous injections) at Week 0 followed by placebo matched to adalimumab (1 subcutaneous injection) at Weeks 1, 3, and 5 and every 2 weeks thereafter through Week 47.
- Adalimumab (ACP): Participants received adalimumab 80 mg (2 subcutaneous injections) at Week 0 and adalimumab 40 mg (1 subcutaneous injection) at Weeks 1, 3, 5 and once every 2 weeks thereafter through Week 47 and placebo matched to guselkumab subcutaneous injection at Weeks 0, 4, 12, 16, 20 and once every 8 weeks thereafter through Week 44.
- Adalimumab Then Guselkumab 100 mg (After ACP): Participants initially randomized to adalimumab entered a washout period after their final dose at Week 47 and crossed over to receive guselkumab 100 mg subcutaneously q8w at Week 52 and thereafter through Week 252. This arm reports safety data for participants that crossed over to guselkumab from adalimumab.
- Guselkumab Combined: All participants who crossed over to receive guselkumab (GUS) 100 mg subcutaneously at Week 16 from placebo group and participants who were randomized to guselkumab 100 mg group at Week 0. Placebo crossover participants were included in the guselkumab column after crossover to guselkumab. Participants that discontinued treatment prematurely were followed up for safety and hence were included in the safety data. Therefore, combined safety results are reported for this arm. This arm reports safety data for guselkumab.
Arm/Group | Placebo (PCP) | Guselkumab 100 mg (PCP) | Adalimumab (PCP) | Placebo Then Guselkumab 100 mg (ACP) | Guselkumab 100 mg (ACP) | Adalimumab (ACP) | Adalimumab Then Guselkumab 100 mg (After ACP) | Guselkumab Combined
Serious Adverse Events (participants affected / at risk) | 3/174 | 8/329 | 6/333 | 5/165 | 8/324 | 10/326 | 34/280 | 79/494
Other Adverse Events (participants affected / at risk) | 51/174 | 101/329 | 98/333 | 67/165 | 134/324 | 137/326 | 193/280 | 307/494
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (PCP) (N=174) | Guselkumab 100 mg (PCP) (N=329) | Adalimumab (PCP) (N=333) | Placebo Then Guselkumab 100 mg (ACP) (N=165) | Guselkumab 100 mg (ACP) (N=324) | Adalimumab (ACP) (N=326) | Adalimumab Then Guselkumab 100 mg (After ACP) (N=280) | Guselkumab Combined (N=494)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aortic Valve Incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus Node Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermoid Cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterocutaneous Fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal Strangulation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess Limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Acute Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 3
Chronic Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ovarian Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia Staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scrotal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Avulsion Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foreign Body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Jaw Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post Procedural Fistula (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural Hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendon Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Human Chorionic Gonadotropin Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lateral Patellar Compression Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meniscal Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Epiglottic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Invasive Papillary Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant Melanoma in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Papillary Cystadenoma Lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Balance Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Idiopathic Partial Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacunar Infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abortion Missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Substance Abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine Polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary Sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythrodermic Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lichen Planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral Artery Stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis Superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (PCP) (N=174) | Guselkumab 100 mg (PCP) (N=329) | Adalimumab (PCP) (N=333) | Placebo Then Guselkumab 100 mg (ACP) (N=165) | Guselkumab 100 mg (ACP) (N=324) | Adalimumab (ACP) (N=326) | Adalimumab Then Guselkumab 100 mg (After ACP) (N=280) | Guselkumab Combined (N=494)
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 4 | 6 | 8 | 4 | 13 | 28
Injection Site Erythema (General disorders) | 1 | 6 | 17 | 3 | 4 | 11 | 7 | 5
Bronchitis (Infections and infestations) | 2 | 2 | 3 | 5 | 4 | 7 | 19 | 23
Gastroenteritis (Infections and infestations) | 2 | 5 | 2 | 3 | 11 | 4 | 14 | 25
Influenza (Infections and infestations) | 0 | 2 | 2 | 1 | 2 | 2 | 16 | 20
Nasopharyngitis (Infections and infestations) | 17 | 30 | 36 | 34 | 65 | 57 | 89 | 148
Pharyngitis (Infections and infestations) | 0 | 0 | 2 | 1 | 5 | 7 | 17 | 18
Sinusitis (Infections and infestations) | 0 | 3 | 1 | 3 | 7 | 6 | 14 | 19
Upper Respiratory Tract Infection (Infections and infestations) | 9 | 25 | 16 | 17 | 31 | 33 | 69 | 107
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 11 | 8 | 2 | 10 | 8 | 26 | 37
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 5 | 1 | 7 | 12 | 22 | 28
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 14 | 12
Headache (Nervous system disorders) | 7 | 14 | 13 | 1 | 7 | 16 | 17 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 6 | 10 | 8 | 20 | 24
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 5 | 7 | 0 | 3 | 6 | 7 | 16
Hypertension (Vascular disorders) | 4 | 10 | 7 | 6 | 5 | 10 | 17 | 40

LIMITATIONS AND CAVEATS:
All participants were on guselkumab after Week 48; therefore, there was no concurrent control group within the study after Week 48.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.